CLINICAL TRIAL: NCT02845661
Title: The Correlation of Narcotrend Index and OAA/S Scale in Monitoring Sedation Level With Different Doses of Dexmedetomidine
Brief Title: Correlation of Narcotrend Index and the Observer's Assessment of Alertness/Sedation (OAA/S) Scale
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, bo xu, associate chief physician, Guangzhou General Hospital of Guangzhou Military Command
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Narcotrend index
Record Dates: First submitted 2016-07-24; First posted 2016-07-27 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Anesthesia
Keywords: Narcotrend index; OAA/S scale; Dexmedetomidine; Sedation
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- group 1 (Experimental): patients in group 1, aged 20~60, were accepted an initial dose of 0.9μg/kg dexmedetomidine over 15 min.
  Interventions: Drug: Dexmedetomidine
- group 2 (Experimental): patients in group 2, aged 20~60, were accepted an initial dose of 1.0μg/kg dexmedetomidine over 15 min.
  Interventions: Drug: Dexmedetomidine
- group 3 (Experimental): patients in group 3, aged 20~60, were accepted an initial dose of 1.1μg/kg dexmedetomidine over 15 min.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — a bolus of dexmedetomidine was administered intravenously 15 min after spinal anesthesia,and the initial dose in group 1 was started from 0.9 µg/kg
  Other Names: Dexmedetomidine 0.9 µg/kg
  Arms: group 1
Drug: Dexmedetomidine — a bolus of dexmedetomidine was administered intravenously 15 min after spinal anesthesia,and the initial dose in group 2 was started from 1.0 µg/kg
  Other Names: Dexmedetomidine 1.0 µg/kg
  Arms: group 2
Drug: Dexmedetomidine — a bolus of dexmedetomidine was administered intravenously 15 min after spinal anesthesia,and the initial dose in group 3 was started from 1.1 µg/kg
  Other Names: Dexmedetomidine 1.1 µg/kg
  Arms: group 3

SUMMARY:
Narcotrend index is a widely used quantitative parameter for evaluating anesthesia and sedation levels.Dexmedetomidine is a novel sedative,providing sedation while patients remain cooperative and can be easily aroused. This study was designed to explore the correlation of Narcotrend index and OAA/S scale in monitoring sedation level with different single- doses of dexmedetomidine intravenously.

DETAILED DESCRIPTION:
60 patients,aged 20～60,American Society of Anesthesiologists (ASA) physical status ⅠorⅡ, scheduled for electively lower limb surgery undergoing combined spinal epidural anesthesia were randomly divided three group. In each group,a bolus of dexmedetomidine was administered intravenously 15 min after spinal anesthesia. The initial dose in group 1, group 2 and group 3 was started from 0.9 µg/kg,1.0 µg/kg and 1.1 µg/kg, respectively. HR、MAP、SpO2、the Observer's Assessment of Alertness/Sedation（OAA/S）scale and the corresponding Narcotrend index were recorded at 5-minute intervals until 30 minutes after administration. The relationship between OAA/S scale and Narcotrend index was analyzed by a Spearman analysis. The cutoff values of Narcotrend index for OAA/S≤2 were obtained by analysis of receiver operating characteristic curves(ROC).

ELIGIBILITY:
Inclusion Criteria:

1. ASA Ⅰ ~ Ⅱ women undergoing Laparoscopic surgery.
2. Written informed consent from the patient or the relatives of the participating patient.
3. BMI:18.0～25 kg/m2

Exclusion Criteria:

1. Mental illness can not match
2. epidural anesthesia contraindicated
3. People who have Slow-type arrhythmias
4. Chronic renal failure
5. Alcohol or drug abuse
6. Already taking gabapentin, pregabalin, benzodiazepin or antidepression drug

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
the correlation coefficient between OAA/S scale and Narcotrend index in group 1 | at 5-minute intervals until 30 minutes after administration
  This study was designed to explore the correlation of Narcotrend index and OAA/S scale in monitoring sedation level with different single- doses of 0.9 μg/kg dexmedetomidine intravenously.
the correlation coefficient between OAA/S scale and Narcotrend index in group 2 | at 5-minute intervals until 30 minutes after administration
  This study was designed to explore the correlation of Narcotrend index and OAA/S scale in monitoring sedation level with different single- doses of 1.0 μg/kg dexmedetomidine intravenously.
the correlation coefficient between OAA/S scale and Narcotrend index in group 3 | at 5-minute intervals until 30 minutes after administration
  This study was designed to explore the correlation of Narcotrend index and OAA/S scale in monitoring sedation level with different single- doses of 1.1 μg/kg dexmedetomidine intravenously.

SECONDARY OUTCOMES:
The calculated cutoff values for OAA/S≤ 2 | at 5-minute intervals until 30 minutes after administration

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Military Region General Hospital, Department of Anesthesiology, Guangzhou, Guangdong, China